CLINICAL TRIAL: NCT06400498
Title: Pragmatic Trial Investigating Surprise Question in End of Life (SeQuEL) Care and the Effect of Prompting Palliative Care Consultation on Provider Referral Rates and Subsequent Outcomes for Hospitalized Adults With Serious Illnesses: End-Stage Liver Disease
Brief Title: Surprise Question in End of Life (SeQuEL) Care and the Effect of Prompting Palliative Care Consultation: End-Stage Liver Disease
Acronym: SeQuEL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Mohana Karlekar, Associate Professor of Medicine, Division of General Internal Medicine and Public Health, MD, FACP, FAAHPM, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 240233
Record Dates: First submitted 2024-05-01; First posted 2024-05-06 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: End-Stage Liver Disease
Keywords: Palliative Care
MeSH Terms: conditions — End Stage Liver Disease

STUDY DESIGN:
Intervention Model Description: This study will be performed as a single center, pragmatic, randomized clinical trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No Palliative Care Consultation Prompt Group (No Intervention): When a patient is randomized to the No Palliative Care Consultation Prompt Group, no prompt will occur. A treating clinician can choose to place or discontinue a palliative care consultation at any time. A patient may choose to request or decline a palliative care consultation at any time.
- Palliative Care Consultation Prompt Group (Active Comparator): When a patient is randomized to the Palliative Care Consultation Prompt Group, a clinical decision support tool in the electronic health record will inform the treating clinician of the patient's serious illness and the results of the Surprise Question and prompt the treating clinician to consider a palliative care consultation. A treating clinician can choose to place or discontinue a palliative care consultation at any time, retaining full autonomy to deliver the appropriate patient care. A patient may choose to request or decline a palliative care consultation at any time.
  Interventions: Behavioral: Prompted Palliative Care Consult

INTERVENTIONS:
Behavioral: Prompted Palliative Care Consult — When a patient is randomized to the Palliative Care Consultation Prompt Group, a clinical decision support tool in the electronic health record will inform the treating clinician of the patient's serious illness and the results of the Surprise Question and prompt the treating clinician to consider a palliative care consultation. If the treating clinician feels a palliative care consultation would be indicated for the patient, the clinical decision support tool will facilitate the placement of a palliative care consultation by the treating clinician. If the treating clinician feels that a palliative care consultation would not be indicated, then the clinical decision support will record a reason it is not indicated.
  Arms: Palliative Care Consultation Prompt Group

SUMMARY:
This is a single center randomized platform trial determining whether prompting consideration of palliative care consultation through the electronic health record impacts the number of palliative consultations placed and hospital-free days among hospitalized adults with End-Stage Liver Disease.

DETAILED DESCRIPTION:
Palliative care is specialized medical care focused on providing patients with relief from the symptoms, pain, and stress of serious illness, regardless of diagnosis, by anticipating, preventing, and treating suffering. The goal is to improve quality of life for both the patient and the patient's family. Palliative care is appropriate at any age and at any stage in a serious illness. It may be provided together with curative treatment, and includes intensive focus on symptom and pain management, psychosocial and spiritual support, and assistance in advance care planning.

There is potential benefit to introducing palliative care earlier in the course of illness for patients with chronic liver disease. For some patients with cirrhosis, palliative care has been shown to improve physical and emotional symptoms. In a recent observational study, it was found that for patients with End-Stage Liver Disease (ESLD) on the waiting list for liver transplant, an early palliative care intervention counteracted the progression of worsening symptoms and significantly improved pruritus, appetite, anxiety, depression, fatigue, and well-being. Moreover, the introduction of palliative care within the care course of patients with decompensated cirrhosis is endorsed by an AASLD (American Association for the Study of Liver Diseases) practice guidance document.

Despite the available evidence regarding the potential benefits of specialized palliative care across multiple serious illnesses, the incorporation of palliative care consultation into clinical practice in many settings is inconsistent and often too late in the clinical trajectory. In an effort to introduce palliative care sooner and more consistently into patients' care pathways, the study team will explore an interruptive provider nudge to prompt palliative care consideration in ESLD. This integrated approach will also help bridge the knowledge gap as to whether systematically prompting palliative care consultation can improve referral rates and outcomes for patients with ESLD.

The processes used to 1) identify hospitalized patients with ESLD, 2) query a provider about their status, and 3) prompt consideration of palliative care consultation are amenable to conduct through the electronic health record. Step 1 will employ phenotyping of clinical and admission characteristics readily extractable from the medical record. Step 2 will utilize the "Surprise Question" as a screening tool for identification of potentially unmet palliative care needs. In previous studies of serious illness, patients for whom consideration of palliative care consultation might be appropriate have used the "Surprise Question", which asks the treating clinician "would you be surprised if this patient died in the next 12 months?" Step 3 will harness the capability to prompt a provider to consider appropriately indicated, complementary, supportive care that may be otherwise underutilized while managing the patient's immediate health crisis.

Given the preliminary evidence that specialist palliative care may improve the quality and quantity of time spent alive and outside of the hospital for patients with serious illness and the incomplete implementation of specialty palliative care in current clinical practice, the study team will evaluate the effect of prompting consideration of palliative care consultation in the electronic health record on provider referral rates to the palliative care service and hospital-free days among hospitalized patients with ESLD.

ELIGIBILITY:
Inclusion Criteria:

* Patient is an adult (age ≥ 18 years).
* Patient is admitted to the study hospital.
* Patient meets phenotype criteria for End-Stage Liver Disease.
* Patient's treating physician, physician associate, or nurse practitioner answers "No" to a prompt in the electronic health record asking, "Would you be surprised if this patient died in the next 12 months?"

Exclusion Criteria:

* Patient is known to have received any VUMC palliative care consultation during the prior 3 months and/or the current admission.
* Patient is known to be a prisoner.
* Patient has received a liver transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2024-08-05 (Actual); Primary Completion 2025-05-05 (Actual); Study Completion 2025-08-05 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with palliative care consults placed within 48 hours after enrollment | 48 hours post-enrollment
  Percentage of patients identified within the EHR identified with palliative care consults.
Hospital-free days by day 90 | 90 days post-enrollment
  The number of calendar days between enrollment and day 90 in which the patient is alive and outside of an acute-care hospital. Days spent at home, at a rehabilitation facility, at a nursing facility, and at an inpatient hospice facility will count as hospital-free.

SECONDARY OUTCOMES:
Survival to day 90 | 90 days post-enrollment
  The number of calendar days in which the patient is alive between enrollment and day 90.

CONTACTS AND LOCATIONS:
Overall Officials: Mohana Karlekar, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported will be made available (including data dictionaries) after de-identification.
Supporting Information: Study Protocol, SAP
Time Frame: The data will become available 3 months following publication of outcomes and will remain available for at least 5 years.
Access Criteria: Data will be made available to researchers who provide a methodologically sound proposal that has been approved by the Vanderbilt Institutional Review Board and the study executive committee.

REFERENCES:
- [Background] Ferrell BR, Twaddle ML, Melnick A, Meier DE. National Consensus Project Clinical Practice Guidelines for Quality Palliative Care Guidelines, 4th Edition. J Palliat Med. 2018 Dec;21(12):1684-1689. doi: 10.1089/jpm.2018.0431. Epub 2018 Sep 4. PMID 30179523
- [Background] Reframing Palliative Care | Messages Matter | On-Demand Webinar.; 2017. https://www.capc.org/events/recorded-webinars/reframing-palliative-care-messages-matter/
- [Background] Radbruch L, De Lima L, Knaul F, Wenk R, Ali Z, Bhatnaghar S, Blanchard C, Bruera E, Buitrago R, Burla C, Callaway M, Munyoro EC, Centeno C, Cleary J, Connor S, Davaasuren O, Downing J, Foley K, Goh C, Gomez-Garcia W, Harding R, Khan QT, Larkin P, Leng M, Luyirika E, Marston J, Moine S, Osman H, Pettus K, Puchalski C, Rajagopal MR, Spence D, Spruijt O, Venkateswaran C, Wee B, Woodruff R, Yong J, Pastrana T. Redefining Palliative Care-A New Consensus-Based Definition. J Pain Symptom Manage. 2020 Oct;60(4):754-764. doi: 10.1016/j.jpainsymman.2020.04.027. Epub 2020 May 6. PMID 32387576
- [Background] Baumann AJ, Wheeler DS, James M, Turner R, Siegel A, Navarro VJ. Benefit of Early Palliative Care Intervention in End-Stage Liver Disease Patients Awaiting Liver Transplantation. J Pain Symptom Manage. 2015 Dec;50(6):882-6.e2. doi: 10.1016/j.jpainsymman.2015.07.014. Epub 2015 Aug 22. PMID 26303186
- [Background] Rogal SS, Hansen L, Patel A, Ufere NN, Verma M, Woodrell CD, Kanwal F. AASLD Practice Guidance: Palliative care and symptom-based management in decompensated cirrhosis. Hepatology. 2022 Sep;76(3):819-853. doi: 10.1002/hep.32378. Epub 2022 Apr 22. No abstract available. PMID 35103995
- [Background] Holden JH, Shamseddeen H, Johnson AW, Byriel B, Subramoney K, Cheng YW, Saito A, Ghabril M, Chalasani N, Sachs GA, Orman ES. Palliative Care and Hospice Referrals in Patients with Decompensated Cirrhosis: What Factors Are Important? J Palliat Med. 2020 Aug;23(8):1066-1075. doi: 10.1089/jpm.2019.0501. Epub 2020 Feb 24. PMID 32091954
- [Background] Woodrell CD, Goldstein NE, Moreno JR, Schiano TD, Schwartz ME, Garrido MM. Inpatient Specialty-Level Palliative Care Is Delivered Late in the Course of Hepatocellular Carcinoma and Associated With Lower Hazard of Hospital Readmission. J Pain Symptom Manage. 2021 May;61(5):940-947.e3. doi: 10.1016/j.jpainsymman.2020.09.040. Epub 2020 Oct 6. PMID 33035651
- [Background] Shinall MC Jr, Karlekar M, Martin S, Gatto CL, Misra S, Chung CY, Porayko MK, Scanga AE, Schneider NJ, Ely EW, Pulley JM, Jerome RN, Dear ML, Conway D, Buie R, Liu D, Lindsell CJ, Bernard GR. COMPASS: A Pilot Trial of an Early Palliative Care Intervention for Patients With End-Stage Liver Disease. J Pain Symptom Manage. 2019 Oct;58(4):614-622.e3. doi: 10.1016/j.jpainsymman.2019.06.023. Epub 2019 Jul 2. PMID 31276810
- [Background] Moroni M, Zocchi D, Bolognesi D, Abernethy A, Rondelli R, Savorani G, Salera M, Dall'Olio FG, Galli G, Biasco G; on behalf of the SUQ-P group. The 'surprise' question in advanced cancer patients: A prospective study among general practitioners. Palliat Med. 2014 Jul;28(7):959-964. doi: 10.1177/0269216314526273. Epub 2014 Mar 24. PMID 24662237
- [Background] Moss AH, Ganjoo J, Sharma S, Gansor J, Senft S, Weaner B, Dalton C, MacKay K, Pellegrino B, Anantharaman P, Schmidt R. Utility of the "surprise" question to identify dialysis patients with high mortality. Clin J Am Soc Nephrol. 2008 Sep;3(5):1379-84. doi: 10.2215/CJN.00940208. Epub 2008 Jul 2. PMID 18596118

DOCUMENTS (2):
  • Study Protocol (2024-07-31): https://cdn.clinicaltrials.gov/large-docs/98/NCT06400498/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-03): https://cdn.clinicaltrials.gov/large-docs/98/NCT06400498/SAP_001.pdf